CLINICAL TRIAL: NCT05698251
Title: Piloting an Intervention Using Single Case Design to Reduce Uncertainty Distress in Those With Long Term Health Conditions
Brief Title: Reducing Uncertainty Distress in Long Term Health Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Northumberland, Tyne and Wear NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sarah Kay, Principle Investigator, Newcastle University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RES-21-015; 21/ES/0063 (Other: East of Scotland Research Ethics Service REC 1); 293383 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2022-12-23; First posted 2023-01-26 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Rheumatic Diseases
Keywords: Uncertainty
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: Single Case Design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reducing uncertainty distress: Psychological therapy intervention (Experimental): Up to 16 sessions of psychological therapy delivered weekly either face to face or via telehealth . Based on empirically grounded models of anxiety/threat, illness uncertainty and intolerance of uncertainty.
  Formulation driven and clinically responsive individualised treatment based on four intervention areas: information management, building safety, reducing overestimation of threat and tolerating uncertainty.
  Interventions: Behavioral: Uncertainty distress model

INTERVENTIONS:
Behavioral: Uncertainty distress model — Psychological therapy intervention based on elements of traditional Cognitive Behaviour Therapy (CBT) for anxiety, illness uncertainty and intolerance of uncertainty.

SUMMARY:
The goal of this pilot intervention study is to develop and test a new psychological therapy model in people with long term health conditions (rheumatic conditions) who are experiencing distress (anxiety or low mood) in relation to the uncertainty that their illness causes.

The main questions the study aims to answer are:

1. Does the new treatment model help participants reduce uncertainty distress associated with their health condition?
2. Is it a practical treatment that can be ran within a hospital setting?
3. Is the treatment acceptable to participants?

Participants will be asked to attend weekly therapy sessions (up to a maximum of 16 sessions) in the hospital or via telehealth. The sessions will be based on the new treatment model and aimed at helping participants reduce uncertainty where they can and learn to live alongside it where it cannot be reduced. The hope is that if participants can better manage uncertainty this will reduce the distress (anxiety or low mood) that they feel.

DETAILED DESCRIPTION:
Uncertainty is a natural part of chronic illness and is typically experienced as aversive for most people. Sources of uncertainty in illness can include living with ambiguous symptoms, unpredictability of flare ups, if/when the illness will worsen and how effective treatment will be. Whilst some real-world uncertainty is inevitable in illness, perceived uncertainty can be exacerbated by inconsistent and/or inadequate health information. High levels of illness uncertainty have been associated with greater emotional distress/mood disturbances, poorer adjustment and reduced quality of life.

Uncertainty management interventions have traditionally focused on reducing uncertainty through information management strategies. These have been shown to be effective in improving patient knowledge of their condition, improve patient-health professionals communication, mood and coping skills. Research into emotional disorders have identified uncertainty as a transdiagnostic source of distress and studies increasing tolerance of uncertainty have been shown to be effective.

To date there is no research combining informational interventions to reduce perceived uncertainty and interventions increasing tolerance of uncertainty in those with chronic health conditions. The aim of this study is pilot a transdiagnostic treatment model combining both elements. The intervention consists of 4 main interventional areas; information management, building safety, addressing overestimation of threat, and tolerating uncertainty. This treatment has the potential to reduce disease distress and burden and potentially reduce health care utilisation if patients are managing their health conditions and associated uncertainty better.

Using single case design this study will look to develop and evaluate the new treatment intervention. The aim is to establish whether his treatment is feasible and acceptable to be delivered within a health care setting.

Up to 6 participants will be recruited from the Rheumatology department within a hospital setting. Participants will be experiencing distress related to the uncertainty of their diagnosed health condition and willing to engage in a psychological treatment to reduce distress.

Treatment will consist of 16 weekly therapy sessions (dependent on clinical need) delivered face to face or via telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Long Term Health Condition (Rheumatic Disease)
* Minimum of 12 months since diagnosis
* Difficulties adjusting to long term health condition
* Willingness to engage with a psychological treatment to manage distress associated with health condition
* Fluent English Speaker

Exclusion Criteria:

* Multiple long term health conditions
* Progressive health conditions
* Experiencing mental health difficulties that might interfere with ability to engage in time limited psychological therapy such as Major Depressive Episode and/or severe and enduring mental health problems, comorbid substance misuse, suicidality
* Diagnosis of Autism Spectrum Disorder (ASD)
* Non- English Speaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in daily diary measures | Daily from baseline to follow up (approximately 24 weeks)
  Idiosyncratic statements regarding uncertainty and distress rated on Likert scale. Minimum score 0, Maximum Score 10. Direction of improved scores are dependent on individual statements.

SECONDARY OUTCOMES:
Changes in Patient Health Questionnaire (PHQ9) score | Baseline (Week 0), start of therapy (Week 2-4 depending on randomisation to baseline length) prior to each therapy session (weekly from weeks 2-4 to approximately weeks 18-20) end of therapy (approximately week 20) and follow up (approximately week 24)
  Depression Questionnaire. Scores range from 0 (minimum) to 27 (maximum). Lower scores indicate better outcome
Changes in Generalised Anxiety Disorder (GAD7) score | Baseline (Week 0), start of therapy (Week 2-4 depending on randomisation to baseline length) prior to each therapy session (weekly from weeks 2-4 to approximately weeks 18-20) end of therapy (approximately week 20) and follow up (approximately week 24)
  Anxiety Questionnaire. Scores range from 0 (minimum) to 21 (maximum). Lower scores indicate better outcome.
Changes in Brief Pain Inventory (BPI score) | At 5 time points: Baseline (Week 0), Start of Treatment (Between week 2- week 4 dependent on randomisation to baseline) , Mid treatment (Approximately week 12), End of treatment (Approximately week 20) and Follow up (Approximately week 24)
  Pain measure. Two subscales pain severity and pain interference. Lower scores indicate better outcome.
Changes in scores on Mishels Illness Uncertainty Scale Community version (MUIS-C) | At 5 time points: Baseline (Week 0), Start of Treatment (Approximately week 4) , Mid treatment (Approximately week 12), End of treatment (Approximately week 20) and Follow up (Approximately week 24)
  Measure of illness uncertainty. Scores from 23 (minimum) to 115 (maximum). Lower scores indicate better outcome.
Changes in scores on Intolerance of Uncertainty Scale (IUS)- short form | At 5 time points: Baseline (Week 0), Start of Treatment (Approximately week 4) , Mid treatment (Approximately week 12), End of treatment (Approximately week 20) and Follow up (Approximately week 24)
  Measure of intolerance of uncertainty. Scores from 12 (minimum) to 60 (maximum). Lower scores indicate better outcome.
Changes in scores on Intolerance of Uncertainty Behaviours in Everyday Life Questionnaire (IUBEL) | At 5 time points: Baseline (Week 0), Start of Treatment (Approximately week 4) , Mid treatment (Approximately week 12), End of treatment (Approximately week 20) and Follow up (Approximately week 24)
  Measure of uncertainty behaviours. Two subscales generic and situational subscales. Scores from 0 (minimum) to 96 (maximum) on each subscale. Lower numbers indicate better outcome.
Changes in scores on International Adjustment Disorder Questionnaire (IADQ) | Pre and post treatment (Week 0 and approximately week 24)
  Measure of adjustment to physical illness. Scores from 0 (minimum) to 40 (maximum). Lower numbers indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Freeston, ProfPsy, Study Director — Newcastle University
Locations (1):
- Royal Victoria Hospital (RVI), Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mishel MH. Reconceptualization of the uncertainty in illness theory. Image J Nurs Sch. 1990 Winter;22(4):256-62. doi: 10.1111/j.1547-5069.1990.tb00225.x. PMID 2292449
- [Background] Freeston M, Tiplady A, Mawn L, Bottesi G, Thwaites S. Towards a model of uncertainty distress in the context of Coronavirus (COVID-19). Cogn Behav Therap. 2020 Jul 7;13:e31. doi: 10.1017/S1754470X2000029X. eCollection 2020. PMID 34191941
- [Background] Kuang, K. (2018). Reconceptualizing uncertainty in illness: commonalities, variations, and the multidimensional nature of uncertainty. Annals of the International Communication Association, 42(3), 181-206.
- [Background] Kuang, K., & Wilson, S. R. (2017). A meta-analysis of uncertainty and information management in illness contexts. Journal of Communication, 67(3), 378-401.
- [Background] Zhang Y. Uncertainty in Illness: Theory Review, Application, and Extension. Oncol Nurs Forum. 2017 Nov 1;44(6):645-649. doi: 10.1188/17.ONF.645-649. PMID 29052657

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT05698251/Prot_SAP_000.pdf